CLINICAL TRIAL: NCT06942546
Title: The Use and Meaning of Wrist Orthosis for Persons With Distal Radius Fracture After Cast Removal
Brief Title: Use and Meaning of Wrist Orthosis After Distal Radius Fracture
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Narhalsan primary care rehabilitation (Unknown); Sjukhusen i vaster (Unknown); Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 257381
Record Dates: First submitted 2020-11-10; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Wrist Fracture; Distal Radius Fracture
Keywords: rehabilitation; wrist orthosis; occupational therapy; everyday occupation
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wrist orthosis — The wrist orthosis referred in this study is two different prefabricated (of the shelf) types; a semi-rigid orthosis in elastic fabric with a volar splint or a short elastic wrist orthosis without a splint. Both ment to be worn when the person use the hand in everyday occupation.

SUMMARY:
The aim of this study is to investigate the use and meaning of wrist orthosis in everyday occupation after cast removal for adults with non-surgical treatment of distal radius fracture.

DETAILED DESCRIPTION:
To be able to do meaningful occupations in everyday life is important for human health and well-being. We use our hands in mostly activities and the hands is also used to interpret and express feelings as a social link to others. A traumatic hand injury, such as a distal radius fracture (DRF), alter the conditions for everyday occupation for the person affected.

DRF affects 25,000 people in Sweden each year. The treatment is either conservative with a plaster cast for approximately four weeks, or surgical. At time for cast removal the fracture is clinical stable, but cannot withstand full load in everyday occupations. Normally the person has difficulties to grip and to use the hand.

The occupational therapist (OT) provide the person with information, training program and often a wrist orthosis. The purpose of the wrist orthosis is to reduce pain, risk of overload of the fracture and to facilitate the use of the hand. The wrist orthosis referred in this study is two different prefabricated (of the shelf) types; a semi-rigid orthosis in elastic fabric with a volar splint or a short elastic wrist orthosis without a splint. Both meant to be worn when the person use the hand in everyday occupation. These wrist orthosis is commonly used in Sweden.

There is a lack research of this kind of wrist orthosis after cast removal for persons with DRF. There are studies of passive treatment orthosis designed to increase movement of the wrist or to reduce pain. Those orthosis is not meant to be worn in everyday occupation. There is however support in research that semi-rigid wrist orthosis i beneficial for persons with rheumatoid arthritis.

Method:

The study has a mixed method design, with a initial quantitative phase with data collection and analysis followed by a qualitative phase with interviews of a sample of the study participants.

After trauma and initial care the person with DRF comes to the hospital for a one week check with/without X-ray. At this point written study information is given to persons meeting the inclusion criteria.

At four weeks after trauma the person with DRF visit an OT to get plaster removal. Treatment as usual (TAU) is given. Then an assessment is made and if the patient meet the inclusion criteria and wish to participate in the study a written informed consent will be obtained. Mobility of the wrist in extension and flexion is measured. The participant is provided with a wrist orthosis and the ordination to use it when needed, where need is described as reducing pain, facilitation of the use of the hand or improved rest för the wrist. A diary and instruction on registration is given. It's to be done approximately one week from cast removal.

At six weeks after trauma a revisit is made. TAU together with collection of the diary. Also there is data collection with patient rated wrist evaluation (PRWE) and measurement of wrist mobility. Information of planned follow-up at Three months after trauma.

At ten weeks after trauma a letter is sent to the participant with a diary and PRWE. The participant is asked to fill in these and bring them to the clinic at revisit.

At twelve weeks after trauma a revisit to the clinic is made. At the visit measure of mobility of the wrist is taken and the diary and PRWE is collected.

At twelve to fourteen weeks after trauma a semi-structured qualitative interview is conducted for a smaller sample of participants. The question areas is about the use and meaning of wrist orthosis in everyday occupation during the time from cast removal till now for the participant.

The following quantitative data will be collected:

* Demographic data: gender, age, fracture site in dominant or not-dominant hand, if the fracture was undisplaced or replaced, amount of energy in violence responsible for the fracture and number of days in plaster. Also professional activity and days of sick-leave and days before return to work.
* Mobility of the wrist in extension and flexion, measured with goniometer.
* The use and benefit of the wrist orthosis is measured with a diary, which is filled in at 5-6 weeks and 10-11 weeks after trauma. It gives data of time with and without wrist orthosis, in which types of occupation wrist orthosis was used and what benefit was experienced.
* Pain and ability to use the affected hand is measured with PRWE.

Qualitative data is collected through semistructured interviews with a smaller sample of participants. The main question will be: "What significance has the wrist orthosis had for you during the time from plaster removal to today?" During the interview the persons diaries is used as a background for reflection.

Inclusions criteria:

Adult with unilateral distal radius fracture treated conservative with plaster for 25-31 days treated at Alingsås hospital and given plaster removal and rehabilitation by occupational therapist in hospital care or primary care in Alingsås.

Exclusion criteria:

* At plaster removal no pain in the wrist and less than 20 degrees decrease of mobility in the wrist in extension/flexion/pronation/supination since they are not deemed to be in need of wrist orthosis.
* Other disease which highly affect pain, joint mobility and/or strength such as rheumatoid arthritis, severe arthritis or neurological disease.
* Not able to communicate in Swedish
* Obvious cognitive impairment

Sample size:

In the planned pilot study 30 participants will be enrolled. Interview will be conducted with 6-10 participants.

ELIGIBILITY:
Inclusion Criteria:

* adults with unilateral distal radius fracture, non-operated, treated with cast for 25-31 Days
* participants shall be treated at Sjukhusen i väster/Alingsås lasarett and get rehabilitation from occupational therapist in hospital rehabilitation clinic or in primary care rehabilitation clinic in Alingsås

Exclusion Criteria:

* At time for decasting are pain free and have less than 20 degrees reduction of ROM in the wrist
* Another disease or injury that affects pain, joint mobility and/or strength such as rheumatoid arthritis or neurological disease.
* Not able to communicate in Swedish, due to self-report Formulas and interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult whit distal radius fracture Treated without surgery, but with casting for 25-31 Days Gets rehabilitation at Sjukhusen i väster/Alingsås lasarett or in Primary care rehabilitation in Alingsås
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Time for use of wrist orthosis | 5-6 weeks after fracture and 12 weeks after fracture
  self-reported values of time with wrist orthosis day-time and during night
Type of activities with wrist orthosis | 5-6 weeks after fracture and 12 weeks after fracture
  Self-reported values of type of activities with wrist orthosis, activities categorized accordingly to Canadian Occupational Performance Measure
Perceived usefulness and value of wrist orthosis in different activities | 5-6 weeks after fracture and 12 weeks after fracture
  self-reported value of usefulness/value in different activities

SECONDARY OUTCOMES:
Type of usefulness of the wrist orthosis | 5-6 weeks after fracture and 12 weeks after fracture
  self-reported types of usefulness
Type of obstacles of the wrist orthosis | 5-6 weeks after fracture and 12 weeks after fracture
  self-reported types of obstacles of the wrist orthosis

OTHER OUTCOMES:
qualitative data of the experiences of usage of wrist orthosis the first time after wrist fracture | at 12-14 weeks after fracture
  content analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Sjukhusen i väster Rehabmottagning Alingsås, Alingsås, Sweden